CLINICAL TRIAL: NCT01438619
Title: Sodium Intake: Research for the Improvement in Measurement Methods and the Effect of Sodium Intake on Cardiovascular Health
Brief Title: Research for the Improvement in Measurement Methods and the Effect of Sodium Intake on Cardiovascular Health
Status: Completed | Type: Observational
Sponsor: DongGuk University (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Professor, DongGuk University
Other Study IDs: 11162KFDA162; 11162KFDA162 (Other Grant/Funding Number: 11162KFDA162)
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Sodium Intake; General Population
Keywords: sodium; blood pressure; pulse wave velocity; random digit dialling

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- representitives of Goyang city: 1. Representative population of Goyang city who were randomly selected by digit dialing (RDD) method
  2. Volunteers who are reside in Goyang city

SUMMARY:
Epidemiological, clinical and animal-experimental evidence shows a direct relationship between dietary sodium intake, blood pressure and cardiovascular event. Diverse questionnaire and 24 hour urinary sodium measurement are used to estimate sodium intake. Complete reflection of eating and cooking habits to the dietary survey method is difficult. Furthermore, the differences of database between countries make it difficult to compare the amount of sodium intake between countries. It is also difficult to consider individual variation of cooking and eating habits. Due to limitations of dietary survey method, WHO recommended 24 hour urinary sodium measurement to estimated sodium intake in the population survey, and many countries are adopting. However, in Korea National Health and Nutrition Examination Survey, only dietary survey method has been used.

The present survey study was designed 1) to test the feasibility of 24 hour urinary sodium measurement for the estimation of sodium intake (including percentage of complete 24 hour urine sample collection) in the population based study; 2) to establish feasible method of 24 hour urinary sodium measurement; 3) to compare 24 hour urinary sodium measurement to the dietary survey method; and 4) to estimate the sodium intake by 24 hour urinary sodium measurement in Goyang city general population (aged 20-70 years).

DETAILED DESCRIPTION:
Measurements: should be performed for 2 days

1. 24 hour urine Na, K and Creatinine, 24 hour urine amount

   1. Calculation of urine completeness index : Creatinine/(21 x Bwt)
   2. Definition of incomplete urine collection: complete index less than 0.7 and loss of urine more than one time or 100 mL
2. 24 hour ambulatory blood pressure

   1. mobile-O-graph (IEM GmbH)
   2. measurement interval: 30 minutes
3. Measurement of peripheral blood pressure : microlife WatchBP office

   1. Sitting position
   2. After 5 minutes resting
   3. Peripheral systolic BP (pSBP), Peripheral diastolic BP (pDBP),
4. Central aortic blood pressure

   1. SphygmoCor (AtCor Medical, Australia)
   2. Central systolic blood pressure
5. Pulse wave velocity

   1. VP2000 (Colin, Japan)
   2. pulse wave velocity (PWV): carotid-femoral Pulse Wave Velocity, heart-femoral Pulse Wave Velocity and brachial-ankle Pulse Wave Velocity
   3. distance measured by tape: distance from suprasternal notch to carotid artery, distance from suprasternal notch to femoral artery
   4. Silent environment
6. Electrocardiography
7. Blood chemistry and complete blood count

   1. Measure at the morning of first day after overnight fasting
   2. complete blood count, blood urea nitrogen/Creatinine, Fasting blood glucose, Total cholesterol, triglyceride, HDL cholesterol

Measurement protocol

1. 1st day

   1. Visit hospital before 9:00 AM after overnight fasting
   2. Sampling of venous blood
   3. start 24 hour urine collection from 9:00 AM (with education for complete collection)
   4. start 24 hour ambulatory blood pressure monitoring, in parallel with 24 hour urine collection
2. 2nd day

   1. Measure central aortic blood pressure
   2. Measure Pulse Wave Velocity
   3. Electrocardiography

ELIGIBILITY:
Inclusion Criteria:

* General population who are reside in Goyang city

Exclusion Criteria:

* Urinary tract disease
* Known chronic kidney disease
* Unable to measure 24 hour ambulatory blood pressure measurement
* Unable to collect 24 hour urine sample
* Pregnancy
* Alcoholics
* Severe liver disease
* Night workers
* Mental retardation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Representative population of Goyang city who were randomly selected by digit dialing (RDD) method
  2. Volunteers who are reside in Goyang city
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Sodium intake in a studied community | Cross-section
  Sodium intake of a community population is measured by 24 hour urinary sodium excretion

SECONDARY OUTCOMES:
The association between 24 hour urinary sodium excretion and ambulatory blood pressure | Cross-sectional

OTHER OUTCOMES:
The relationship between ambulatory blood pressure variability and arterial stiffness | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, MD, PhD, Principal Investigator — Clinical Trial Center, Dongguk University Ilsan Hospital
Locations (1):
- Clinical Trial Center, Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea